CLINICAL TRIAL: NCT03768349
Title: PSMA and C-11 Choline PET in Patients With Biochemical Recurrence of Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Val Lowe, Prinicpal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-006159; NCI-2019-07001 (Registry Identifier: Clinical Trials Reporting Program (CTRP)); 18-006159 (Other: Mayo Clinic Institutional Review Board); MC1952 (Other: Mayo Clinic); NCT04144010 (obsolete NCT alias)
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PET/CT; PSMA; C-11 Choline
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PET/CT Ga-68 PSMA (Experimental): Ga-68 labeled PSMA-11 (or PSMA-HBED-CC) PET/CT
  Interventions: Drug: Ga-68 PSMA11
- PET/CT F-18 Labeled PSMA 1007 (Experimental): F-18 Labeled PSMA 1007 PET/CT
  Interventions: Drug: F-18 PSMA 1007

INTERVENTIONS:
Drug: Ga-68 PSMA11 — Ga-68 PSMA11 PET/CT for detection of tumor location
  Arms: PET/CT Ga-68 PSMA
Drug: F-18 PSMA 1007 — F-18 PSMA 1007 PET/CT for detection of tumor location
  Arms: PET/CT F-18 Labeled PSMA 1007

SUMMARY:
Imaging and staging of prostate cancer is critical for surgical and treatment planning. In this protocol we will image patients with suspected metastatic prostate cancer using 11C-Choline PET and Gallium-68 labeled HBED-CC PSMA (more commonly called 68Ga-PSMA-11) or F-18 labeled PSMA 1007 in order to demonstrate their utility in detecting prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological proven prostate adenocarcinoma.
2. Rising PSA after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy).

   a. Post radical prostatectomy (RP) - with or without radiation. i. PSA greater than or equal to 0.2 ng/mL measured more than 12 weeks after RP. ii. > 3 months post-surgery b. Post-radiation therapy ASTRO-Phoenix consensus definition c. May or may not be castrate resistant (list prior therapies)
3. Karnofsky performance status of 50 (or ECOG/WHO equivalent).
4. CT or as part of the PET study or performed within one month of PSMA PET.
5. Age > 18.
6. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Undergoing investigational therapy for prostate cancer.
2. Other ongoing treatments for prostate cancer including radiation therapy, chemotherapy or androgen deprivation. Androgen deprivation within the last 4 months excluding finasteride, dutasteride or other 5 alpha reductase inhibitors (excluding castrate resistant subjects).
3. Unable to lie flat, still or tolerate a PET scan.
4. Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.
5. Contraindication to furosemide administration including prior allergy or adverse reaction to furosemide or sulfa drugs. (Note: This exclusion criteria can be removed if Furosemide is omitted as part of the PET imaging protocol if a second-generation scatter correction is available for the used PET device).
6. Absence of PSA and total testosterone tests within 4 weeks.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Tumor Detection on PET/CT | 12 Months post PET/CT
  Positive predictive value on a per-patient and per-region-basis of PSMA and C-11 choline PET/CT for detection of tumor location confirmed by histopathology/biopsy or conventional imaging follow-up.

SECONDARY OUTCOMES:
Impact of PSMA and C-11 choline PET on clinical management | 12 Months
  Descriptive statistics will be used to evaluate the impact of PSMA and C-11 choline PET on clinical management
Incidence of adverse events attributable to PSMA | 12 Months
  Adverse events will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Val Lowe, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD data from this trial will be available to other researchers that will collate similar data from multiple sites to provide data to the FDA.
Supporting Information: Study Protocol, CSR
Time Frame: After completion of the trial and IPD will be available for 2 years.
Access Criteria: Researchers collating data from multiple sites for submission to the FDA will be provided access to the IPD.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials